CLINICAL TRIAL: NCT00909545
Title: A Pilot Phase II Double-Blind, Placebo-Controlled, Tolerability and Dosage Finding Study of Isradipine CR as a Disease Modifying Agent in Patients With Early Parkinson Disease
Brief Title: Safety, Tolerability and Efficacy Assessment of Dynacirc CR in Parkinson Disease
Acronym: STEADY-PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); Northwestern University Dixon Fund (Unknown); The Parkinson Study Group (Network)
Responsible Party: Principal Investigator, Tanya Simuni, Prinicpal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTCC Protocol #124
Record Dates: First submitted 2009-05-26; First posted 2009-05-28 (Estimated); Results first posted 2013-04-17 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Parkinson Disease
Keywords: Early Parkinson disease
MeSH Terms: conditions — Parkinson Disease | interventions — Isradipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Isradipine CR 5mg (Active Comparator): Isradipine CR 5mg/day
  Interventions: Drug: Isradipine CR 5mg
- Isradipine CR 10mg (Active Comparator): Isradipine CR 10mg/day
  Interventions: Drug: Isradipine CR 10mg
- Isradipine CR 20mg (Active Comparator): Isradipine CR 20mg/day
  Interventions: Drug: Isradipine CR 20mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isradipine CR 5mg — 5mg dose: 1 Dynacirc CR 5mg tablet, 3 tablets placebo once daily
  Other Names: Isradipine CR; Dynacirc CR
  Arms: Isradipine CR 5mg
Drug: Isradipine CR 10mg — 10mg dose: 2 Dynacirc CR 5mg tablets, 2 tablets placebo once daily
  Other Names: Isradipine CR; Dynacirc CR
  Arms: Isradipine CR 10mg
Drug: Isradipine CR 20mg — 20mg dose: 4 Dynacirc CR 5mg tablets once daily
  Other Names: Isradipine CR; Dynacirc CR
  Arms: Isradipine CR 20mg
Drug: Placebo — 4 Placebo to Match (PTM) tablets once daily
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to establish a dosage of isradipine CR that is tolerable and demonstrates preliminary efficacy for utilization in future pivotal efficacy studies.

DETAILED DESCRIPTION:
There is solid scientific rational and preclinical data supporting a clinical trial of isradipine CR as a potential disease modifying agent in early PD. Human pharmacokinetic data demonstrate that it is feasible to achieve the serum concentrations in humans that were neuroprotective in preclinical models with the FDA approved dosage range. Pilot data demonstrate acceptable tolerability of isradipine CR in the PD population. Tolerability is inversely proportional to the dosage dependent. Considering that tolerability of isradipine CR is inversely proportional to the dosage exposure, it is essential to proceed with the dose selection tolerability study in preparation for the future efficacy trials.

The tolerability, defined as the ability to complete the study, of three dosages of isradipine CR relative to placebo in subjects with early Parkinson's disease will be examined first. The dosage that is tolerable and demonstrates preliminary efficacy will be evaluated further in the future pivotal efficacy studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with early idiopathic PD. If tremor is not present, subjects must have unilateral onset and persistent asymmetry of the symptoms.
* Be over 30 years old at the time of diagnosis of PD.
* Hoehn & Yahr stage is less than or equal to 2.5.
* Currently not receiving dopaminergic therapy and not projected to require dopaminergic therapy for at least 6 months from enrollment.
* Use of MAO-B inhibitors (rasagiline, selegiline), amantadine, or anticholinergics will be allowed. The dosage has to be stable for 3 months prior to baseline visit and throughout the duration of the study.

Exclusion Criteria:

* Subjects with a diagnosis of an atypical Parkinsonism
* Subjects unwilling or unable to give informed consent
* Use of CoQ10 at a dosage >600mg daily or use of creatine >5 grams daily within the 60 days prior to randomization
* Exposure to dopaminergic PD therapy within 60 days prior to enrollment or for 3 months or more at any point in the past
* History of clinically significant orthostatic hypotension or presence of orthostatic hypotension at the screening visit defined as > 20 mmHg change in systolic BP and >10mm change in diastolic BP after 2 min of standing, or baseline BP <90/60
* History of congestive heart failure
* History of bradycardia defined as heart rate <55
* Presence of 2nd or 3rd degree atrioventricular block or other significant ECG abnormalities that in the investigator's opinion would compromise participation in study
* Clinically significant abnormalities in the Screening Visit laboratory studies or electrocardiogram.
* Presence of other known medical or psychiatric comorbidity that in the investigator's opinion would compromise participation in the study
* Prior exposure to isradipine or other calcium channel blockers within 6 months of baseline
* Subjects with history of hypertension treated with a maximum of 2 other antihypertensive agents will be allowed provided that the doses of concomitant anti HTN therapy can be reduced/adjusted during the study based on the BP readings in consultation with the subject's primary care physician or cardiologist.
* Use of grapefruit juice, Ginkgo biloba, St. John's wart and/or ginseng will be prohibited during the study (as they interfere with the metabolism of isradipine).
* Presence of cognitive dysfunction defined by a Mini Mental Status Exam ( MMSE) score < 26 at screening
* Subjects with clinically significant depression as determined by a Beck Depression Inventory (BDI) score >15 at screening
* History of exposure to typical or atypical antipsychotics or other dopamine blocking agents within 6 months prior to enrollment
* Subjects have to be on a stable regimen of central nervous system acting medications (benzodiazepines, antidepressants, hypnotics) for 30 days prior to enrollment
* Lactating women or women of childbearing potential who are not surgically sterilized have to use a reliable measure of contraception and have a negative serum pregnancy test at screening
* Participation in other investigational drug trials within 30 days prior to screening
* History of brain surgery for PD

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Simuni, MS, Study Chair — Northwestern University
Locations (20):
- United States (18):
  - Parkinson Institute, Sunnyvale, California
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - University of South Flordia, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Pacific Health Institute, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Boston University, Boston, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Park Nicolet Clinic, Golden Valley, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
- Canada (2):
  - Ottowa Hospital Civic Site, Ottawa, Ontario
  - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Background] Parkinson Study Group. Effects of tocopherol and deprenyl on the progression of disability in early Parkinson's disease. N Engl J Med. 1993 Jan 21;328(3):176-83. doi: 10.1056/NEJM199301213280305. PMID 8417384
- [Background] Parkinson Study Group. Dopamine transporter brain imaging to assess the effects of pramipexole vs levodopa on Parkinson disease progression. JAMA. 2002 Apr 3;287(13):1653-61. doi: 10.1001/jama.287.13.1653. PMID 11926889
- [Background] Parkinson Study Group. A controlled, randomized, delayed-start study of rasagiline in early Parkinson disease. Arch Neurol. 2004 Apr;61(4):561-6. doi: 10.1001/archneur.61.4.561. PMID 15096406
- [Background] NINDS NET-PD Investigators. A randomized, double-blind, futility clinical trial of creatine and minocycline in early Parkinson disease. Neurology. 2006 Mar 14;66(5):664-71. doi: 10.1212/01.wnl.0000201252.57661.e1. Epub 2006 Feb 15. PMID 16481597
- [Background] NINDS NET-PD Investigators. A randomized clinical trial of coenzyme Q10 and GPI-1485 in early Parkinson disease. Neurology. 2007 Jan 2;68(1):20-8. doi: 10.1212/01.wnl.0000250355.28474.8e. PMID 17200487
- [Background] Becker C, Jick SS, Meier CR. Use of antihypertensives and the risk of Parkinson disease. Neurology. 2008 Apr 15;70(16 Pt 2):1438-44. doi: 10.1212/01.wnl.0000303818.38960.44. Epub 2008 Feb 6. PMID 18256367
- [Background] Braak H, Ghebremedhin E, Rub U, Bratzke H, Del Tredici K. Stages in the development of Parkinson's disease-related pathology. Cell Tissue Res. 2004 Oct;318(1):121-34. doi: 10.1007/s00441-004-0956-9. Epub 2004 Aug 24. PMID 15338272
- [Background] Chan CS, Guzman JN, Ilijic E, Mercer JN, Rick C, Tkatch T, Meredith GE, Surmeier DJ. 'Rejuvenation' protects neurons in mouse models of Parkinson's disease. Nature. 2007 Jun 28;447(7148):1081-6. doi: 10.1038/nature05865. Epub 2007 Jun 10. PMID 17558391
- [Background] Christensen HR, Antonsen K, Simonsen K, Lindekaer A, Bonde J, Angelo HR, Kampmann JP. Bioavailability and pharmacokinetics of isradipine after oral and intravenous administration: half-life shorter than expected? Pharmacol Toxicol. 2000 Apr;86(4):178-82. doi: 10.1034/j.1600-0773.2000.d01-32.x. PMID 10815751
- [Background] de Lau LM, Breteler MM. Epidemiology of Parkinson's disease. Lancet Neurol. 2006 Jun;5(6):525-35. doi: 10.1016/S1474-4422(06)70471-9. PMID 16713924
- [Background] Dodel RC, Singer M, Kohne-Volland R, Szucs T, Rathay B, Scholz E, Oertel WH. The economic impact of Parkinson's disease. An estimation based on a 3-month prospective analysis. Pharmacoeconomics. 1998 Sep;14(3):299-312. doi: 10.2165/00019053-199814030-00006. PMID 10186468
- [Background] Dorsey ER, Constantinescu R, Thompson JP, Biglan KM, Holloway RG, Kieburtz K, Marshall FJ, Ravina BM, Schifitto G, Siderowf A, Tanner CM. Projected number of people with Parkinson disease in the most populous nations, 2005 through 2030. Neurology. 2007 Jan 30;68(5):384-6. doi: 10.1212/01.wnl.0000247740.47667.03. Epub 2006 Nov 2. PMID 17082464
- [Background] Elm JJ, Goetz CG, Ravina B, Shannon K, Wooten GF, Tanner CM, Palesch YY, Huang P, Guimaraes P, Kamp C, Tilley BC, Kieburtz K; NET-PD Investigators. A responsive outcome for Parkinson's disease neuroprotection futility studies. Ann Neurol. 2005 Feb;57(2):197-203. doi: 10.1002/ana.20361. PMID 15668964
- [Background] Fahn S, Oakes D, Shoulson I, Kieburtz K, Rudolph A, Lang A, Olanow CW, Tanner C, Marek K; Parkinson Study Group. Levodopa and the progression of Parkinson's disease. N Engl J Med. 2004 Dec 9;351(24):2498-508. doi: 10.1056/NEJMoa033447. PMID 15590952
- [Background] Gill DJ, Freshman A, Blender JA, Ravina B. The Montreal cognitive assessment as a screening tool for cognitive impairment in Parkinson's disease. Mov Disord. 2008 May 15;23(7):1043-1046. doi: 10.1002/mds.22017. PMID 18381646
- [Background] Goetz CG, LeWitt PA, Weidenman M. Standardized training tools for the UPDRS activities of daily living scale: newly available teaching program. Mov Disord. 2003 Dec;18(12):1455-8. doi: 10.1002/mds.10591. PMID 14673881
- [Background] Goetz CG, Stebbins GT, Chmura TA, Fahn S, Klawans HL, Marsden CD. Teaching tape for the motor section of the unified Parkinson's disease rating scale. Mov Disord. 1995 May;10(3):263-6. doi: 10.1002/mds.870100305. PMID 7544438
- [Background] Huse DM, Schulman K, Orsini L, Castelli-Haley J, Kennedy S, Lenhart G. Burden of illness in Parkinson's disease. Mov Disord. 2005 Nov;20(11):1449-54. doi: 10.1002/mds.20609. PMID 16007641
- [Background] Jankovic J, Hunter C. A double-blind, placebo-controlled and longitudinal study of riluzole in early Parkinson's disease. Parkinsonism Relat Disord. 2002 Mar;8(4):271-6. doi: 10.1016/s1353-8020(01)00040-2. PMID 12039422
- [Background] Johnson BA, Javors MA, Lam YW, Wells LT, Tiouririne M, Roache JD, Ait-Daoud N, Lawson K. Kinetic and cardiovascular comparison of immediate-release isradipine and sustained-release isradipine among non-treatment-seeking, cocaine-dependent individuals. Prog Neuropsychopharmacol Biol Psychiatry. 2005 Jan;29(1):15-20. doi: 10.1016/j.pnpbp.2004.08.014. Epub 2004 Nov 11. PMID 15610940
- [Background] Kupsch A, Sautter J, Schwarz J, Riederer P, Gerlach M, Oertel WH. 1-Methyl-4-phenyl-1,2,3,6-tetrahydropyridine-induced neurotoxicity in non-human primates is antagonized by pretreatment with nimodipine at the nigral, but not at the striatal level. Brain Res. 1996 Nov 25;741(1-2):185-96. doi: 10.1016/s0006-8993(96)00917-1. PMID 9001722
- [Background] Leentjens AF, Verhey FR, Luijckx GJ, Troost J. The validity of the Beck Depression Inventory as a screening and diagnostic instrument for depression in patients with Parkinson's disease. Mov Disord. 2000 Nov;15(6):1221-4. doi: 10.1002/1531-8257(200011)15:63.0.co;2-h. PMID 11104209
- [Background] Levy G, Kaufmann P, Buchsbaum R, Montes J, Barsdorf A, Arbing R, Battista V, Zhou X, Mitsumoto H, Levin B, Thompson JL. A two-stage design for a phase II clinical trial of coenzyme Q10 in ALS. Neurology. 2006 Mar 14;66(5):660-3. doi: 10.1212/01.wnl.0000201182.60750.66. PMID 16534103
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Olanow CW, Watts RL, Koller WC. An algorithm (decision tree) for the management of Parkinson's disease (2001): treatment guidelines. Neurology. 2001 Jun;56(11 Suppl 5):S1-S88. doi: 10.1212/wnl.56.suppl_5.s1. No abstract available. PMID 11402154
- [Background] Peto V, Jenkinson C, Fitzpatrick R, Greenhall R. The development and validation of a short measure of functioning and well being for individuals with Parkinson's disease. Qual Life Res. 1995 Jun;4(3):241-8. doi: 10.1007/BF02260863. PMID 7613534
- [Background] Richards M, Marder K, Cote L, Mayeux R. Interrater reliability of the Unified Parkinson's Disease Rating Scale motor examination. Mov Disord. 1994 Jan;9(1):89-91. doi: 10.1002/mds.870090114. PMID 8139610
- [Background] Shults CW, Oakes D, Kieburtz K, Beal MF, Haas R, Plumb S, Juncos JL, Nutt J, Shoulson I, Carter J, Kompoliti K, Perlmutter JS, Reich S, Stern M, Watts RL, Kurlan R, Molho E, Harrison M, Lew M; Parkinson Study Group. Effects of coenzyme Q10 in early Parkinson disease: evidence of slowing of the functional decline. Arch Neurol. 2002 Oct;59(10):1541-50. doi: 10.1001/archneur.59.10.1541. PMID 12374491
- [Background] Simuni T, Borushko E, Avram MJ, Miskevics S, Martel A, Zadikoff C, Videnovic A, Weaver FM, Williams K, Surmeier DJ. Tolerability of isradipine in early Parkinson's disease: a pilot dose escalation study. Mov Disord. 2010 Dec 15;25(16):2863-6. doi: 10.1002/mds.23308. PMID 20818667
- [Background] Striessnig J, Koschak A, Sinnegger-Brauns MJ, Hetzenauer A, Nguyen NK, Busquet P, Pelster G, Singewald N. Role of voltage-gated L-type Ca2+ channel isoforms for brain function. Biochem Soc Trans. 2006 Nov;34(Pt 5):903-9. doi: 10.1042/BST0340903. PMID 17052224
- [Background] Suchowersky O, Gronseth G, Perlmutter J, Reich S, Zesiewicz T, Weiner WJ; Quality Standards Subcommittee of the American Academy of Neurology. Practice Parameter: neuroprotective strategies and alternative therapies for Parkinson disease (an evidence-based review): report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2006 Apr 11;66(7):976-82. doi: 10.1212/01.wnl.0000206363.57955.1b. PMID 16606908
- [Background] Twelves D, Perkins KS, Counsell C. Systematic review of incidence studies of Parkinson's disease. Mov Disord. 2003 Jan;18(1):19-31. doi: 10.1002/mds.10305. PMID 12518297
- [Background] Urien S, Pinquier JL, Paquette B, Chaumet-Riffaud P, Kiechel JR, Tillement JP. Effect of the binding of isradipine and darodipine to different plasma proteins on their transfer through the rat blood-brain barrier. Drug binding to lipoproteins does not limit the transfer of drug. J Pharmacol Exp Ther. 1987 Jul;242(1):349-53. PMID 2956411
- [Background] Whone AL, Watts RL, Stoessl AJ, Davis M, Reske S, Nahmias C, Lang AE, Rascol O, Ribeiro MJ, Remy P, Poewe WH, Hauser RA, Brooks DJ; REAL-PET Study Group. Slower progression of Parkinson's disease with ropinirole versus levodopa: The REAL-PET study. Ann Neurol. 2003 Jul;54(1):93-101. doi: 10.1002/ana.10609. PMID 12838524
- [Background] Zadikoff C, Fox SH, Tang-Wai DF, Thomsen T, de Bie RM, Wadia P, Miyasaki J, Duff-Canning S, Lang AE, Marras C. A comparison of the mini mental state exam to the Montreal cognitive assessment in identifying cognitive deficits in Parkinson's disease. Mov Disord. 2008 Jan 30;23(2):297-9. doi: 10.1002/mds.21837. PMID 18044697

RESULTS

PARTICIPANT FLOW:
Groups:
- Isradipine CR 5mg/Day: 1 Dynacirc CR 5mg tablet, 3 tablets placebo once daily
- Isradipine CR 10mg/Day: 2 Dynacirc CR 5mg tablets, 2 tablets placebo once daily
- Isradipine CR 15-20mg/Day: 3-4 Dynacirc CR 5mg tablets once daily
Period: Overall Study
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 15-20mg/Day
Started | 26 | 23 | 26 | 24
Completed | 25 | 22 | 25 | 19
Not Completed | 1 | 1 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Isradipine CR 20mg/Day: 4 Dynacirc CR 5mg tablets once daily
- Total: Total of all reporting groups
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day | Total
Number analyzed (Participants) | 26 | 23 | 26 | 24 | 99
Age Continuous [Mean (Standard Deviation); unit: years] | 60.2 (10.1) | 57.7 (8.3) | 58.5 (11.6) | 59.8 (8.9) | 59.1 (9.8)
Age, Customized [Number; unit: participants]
  Between 30 and 65 years | 17 | 18 | 18 | 19 | 72
  >=65 years | 9 | 5 | 8 | 5 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 9 | 8 | 30
  Male | 21 | 15 | 17 | 16 | 69
Race/Ethnicity, Customized [Number; unit: participants]
  White | 25 | 22 | 22 | 22 | 91
  Other race | 1 | 1 | 4 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 24 | 21 | 24 | 21 | 90
  Canada | 2 | 2 | 2 | 3 | 9
Unified Parkinson's Disease Rating Scale (UPDRS) Total [Mean (Standard Deviation); unit: Unit of UPDRS scales] — Higher score indicates more severe disability.
  Unit of UPDRS scales | 25.46 (9.39) | 26.43 (9.69) | 23.65 (9.97) | 24.67 (10.77) | 25.0 (9.9)
Unified Parkinson's Disease Rating Scale (UPDRS) Mental [Mean (Standard Deviation); unit: Unit of UPDRS scales] — Higher score indicates more severe disability.
  Unit of UPDRS scales | 0.65 (1.06) | 1.30 (1.79) | 0.65 (0.98) | 0.96 (1.12) | 0.9 (1.3)
Unified Parkinson's Disease Rating Scale (UPDRS) Activities of Daily Living (ADL) [Mean (Standard Deviation); unit: Unit of UPDRS scales] — Higher score indicates more severe disability.
  Unit of UPDRS scales | 5.85 (2.98) | 5.83 (3.02) | 6.15 (3.03) | 6.58 (3.03) | 6.1 (3.0)
Unified Parkinson's Disease Rating Scale (UPDRS) Motor [Mean (Standard Deviation); unit: Unit of UPDRS scales] — Higher score indicates more severe disability.
  Unit of UPDRS scales | 18.96 (7.27) | 19.30 (8.02) | 16.85 (7.88) | 17.13 (8.26) | 18.0 (7.8)
Hoehn & Yahr Scale [Number; unit: Participants] — Higher stage indicates more severe disability.
  Participants
    H/Y Stage: 1 | 7 | 4 | 8 | 11 | 30
    H/Y Stage: 1.5 | 2 | 3 | 0 | 1 | 6
    H/Y Stage: 2 | 16 | 16 | 18 | 11 | 61
    H/Y Stage: 2.5 | 1 | 0 | 0 | 1 | 2
Modified Schwab & England Independence Scale [Mean (Standard Deviation); unit: Percentage scale] — Higher score indicates higher independence.
  Percentage scale | 93.08 (5.11) | 93.48 (4.632) | 93.08 (5.11) | 91.04 (5.10) | 92.0 (5.0)
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: Unit of MoCA] — Lower score indicates more severe disability.
  Unit of MoCA | 26.96 (2.58) | 27.96 (1.97) | 26.92 (2.36) | 27.79 (1.89) | 27.4 (2.2)
PD Qualify of Life Scale [Mean (Standard Deviation); unit: Unit of PDQ-39] — Higher score indicates higher disability.
  Unit of PDQ-39 | 10.28 (8.55) | 9.69 (6.88) | 8.39 (5.82) | 10.45 (8.06) | 9.7 (2.3)
Vital Signs: Systolic [Mean (Standard Deviation); unit: mm Hg]
  Standing | 130.0 (18.12) | 127.3 (17.03) | 130.4 (17.76) | 125.8 (11.96) | 128.4 (16.3)
  Supine | 130.9 (16.04) | 128.5 (13.60) | 131.3 (19.00) | 129.1 (13.69) | 130.0 (15.6)
Vital Signs: Diastolic [Mean (Standard Deviation); unit: mm Hg]
  Standing | 83.73 (12.74) | 84.43 (12.22) | 80.04 (9.73) | 81.29 (11.02) | 82.3 (11.4)
  Supine | 80.69 (11.34) | 79.22 (9.50) | 76.88 (10.95) | 79.63 (10.43) | 79.1 (10.5)
Vital Signs: Pulse [Mean (Standard Deviation); unit: Beats per minute]
  Standing | 72.92 (11.90) | 77.35 (10.70) | 75.50 (12.27) | 72.33 (11.43) | 74.5 (11.6)
  Supine | 68.00 (10.63) | 67.43 (10.28) | 67.08 (8.39) | 66.33 (9.71) | 67.2 (9.6)

OUTCOME MEASURES:

1. Secondary Outcome: Efficacy: Change in Unified Parkinson's Disease Rating Scale (UPDRS)
Description: Outcome is defined as change in total Unified Parkinson's Disease Rating Scale (UPDRS) between the baseline visit and month 12 or the time to require dopaminergic therapy (last visit before subject goes on dopaminergic therapy), whichever occurs first. The UPDRS score has 4 components. Part I assesses mentation; Part II assesses activities of daily living; Part III assesses motor abilities; Part IV assesses complications of therapy. A total of 44 items are included in Parts I-III. Each item will receive a score ranging from 0 to 4 where 0 represents the absence of impairment and 4 represents the highest degree of impairment. Part IV contains 11 items, 4 of these items are scored 0-4 in the same manner, and 7 are scored 0-1, with 0 indicating the absence of impairment and 1 indicating the presence of impairment. Total UPDRS score represents the sum of these items in Parts I-IV. A total of 199 points are possible. 199 represents the worst (total) disability), 0--no disability.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Population: Participants are 99 subjects with early Parkinson disease not requiring dopaminergic therapy.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 15-20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
Scores on a scale | 7.40 (1.39) | 7.44 (1.48) | 6.30 (1.39) | 5.40 (1.45)
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; Change in UPDRS total score of Isradipine CR 5mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.9834, ANCOVA — P-values for efficacy outcomes will be one-sided test with alpha = 0.05; Analysis of covariance is used, with terms representing assigned treatment group and baseline value of the measure in the model; Mean Difference (Net) = 0.04, 95% CI 2-sided [-3.99 to 4.07], Standard Error of Mean 2.03 — Least square mean(standard error) and 95% confidence intervals of the difference between Isradipine CR 5mg and placebo groups is estimated
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; Change in UPDRS total score of Isradipine CR 10mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.5761, ANCOVA — P-values for efficacy outcomes will be one-sided test with alpha = 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.10, 95% CI 2-sided [-5.01 to 2.80], Standard Error of Mean 1.97 — Least square mean(standard error) and 95% confidence intervals of the difference between Isradipine CR 10mg and placebo groups is estimated
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 15-20mg/Day; Change in UPDRS total score of Isradipine CR 20mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.322, ANCOVA — P-values for efficacy outcomes will be one-sided test with alpha = 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -2.00, 95% CI 2-sided [-5.98 to 1.99], Standard Error of Mean 2.01 — Least square mean(standard error) and 95% confidence intervals of the difference between Isradipine CR 20mg and placebo groups is estimated

2. Primary Outcome: Tolerability of the Three Dosages(5mg, 10mg and 20mg) of Isradipine CR.
Description: Tolerability will be judged by the proportion of subjects enrolled in a dosage group able to complete the 12 month study or to the time of initiation of dopaminergic therapy on their original assigned dosage. Tolerability of each active arm will be compared to placebo group.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 25 | 19 | 19 | 9
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; The tolerability of 5mg/day dosage of isradipine CR will be compared with that of the placebo group using one-sided Fisher's exact tests. No adjustment will be made for multiple comparisons in these analyses; Test type: Superiority or Other; p = 0.1383, Fisher Exact; Odds Ratio (OR) = 0.19, 95% CI 2-sided [0.0196 to 1.8411], Standard Error of Mean 1.1587
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; The tolerability of 10mg/day dosage of isradipine CR will be compared with that of the placebo group using one-sided Fisher's exact tests. No adjustment will be made for multiple comparisons in these analyses; Test type: Superiority or Other; p = 0.0248, Fisher Exact; Odds Ratio (OR) = 0.1086, 95% CI 2-sided [0.0123 to 0.9591], Standard Error of Mean 0.1114
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; The tolerability of 20mg/day dosage of isradipine CR will be compared with that of the placebo group using one-sided Fisher's exact tests. No adjustment will be made for multiple comparisons in these analyses; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Odds Ratio (OR) = 0.024, 95% CI 2-sided [0.0028 to 0.2087], Standard Error of Mean 1.1035

3. Secondary Outcome: Efficacy: Change in Mental Subscales of the Unified Parkinson's Disease Rating Scale
Description: The outcome is defined as change in Mental subscale of Unified Parkinson's Disease Rating Scale(UPDRS Part I) between the baseline visit and month 12 or the time of sufficient disability to require dopaminergic therapy. UPDRS Part I: Mentation, behavior and mood, consisting of 4 questions answered on a 0-4 point scale where 0 represents the absence of impairment and 4 represents the highest degree of impairment. Total score represents the sum of these 4 questions. A greater increase in score indicates a greater increase in disability. A total of 16 points are possible. 16 represents the worst (total) disability), 0--no disability.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Population: All participants were used in primary and secondary outcome analyses
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
units on a scale | 0.30 (0.26) | 0.76 (0.28) | 0.30 (0.26) | 0.03 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; Change in Mental UPDRS subscale of Isradipine CR 5mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.2324, ANCOVA; Mean Difference (Net) = 0.46, 95% CI 2-sided [-0.30 to 1.22], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; Change in Mental UPDRS subscale of Isradipine CR 10mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 1, ANCOVA; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.73 to 0.73], Standard Error of Mean 0.37
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; Change in Mental UPDRS subscale of Isradipine CR 20mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.4675, ANCOVA; Mean Difference (Net) = -0.27, 95% CI 2-sided [-1.02 to 0.47], Standard Error of Mean 0.37

4. Secondary Outcome: Efficacy: Change in Activities of Daily Living(ADL) Subscale of the Unified Parkinson's Disease Rating Scale
Description: The outcome is defined as change in ADL subscale of the Unified Parkinson's Disease Rating Scale(UPDRS Part II) between the baseline visit and month 12 or the time of sufficient disability to require dopaminergic therapy. UPDRS Part II: Activities of Daily Living in the week prior to the designated visit, consisting of 13 questions answered on a 0-4 point scale where 0 represents the absence of impairment and 4 represents the highest degree of impairment. Total Part II score represents the sum of these 13 questions. A greater increase in score indicates a greater increase in disability. A total of 52 points are possible. 52 represents the worst (total) disability), 0--no disability
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Population: All participants were included in the primary and secondary outcome analyses
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
units on a scale | 2.60 (0.56) | 3.20 (0.60) | 2.09 (0.56) | 1.86 (0.59)
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; Change in ADL UPDRS subscale of Isradipine CR 5mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.4648, ANCOVA; Mean Difference (Net) = 0.60, 95% CI 2-sided [-1.03 to 2.23], Standard Error of Mean 0.82
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; Change in ADL UPDRS subscale of Isradipine CR 10mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.525, ANCOVA; Mean Difference (Net) = -0.51, 95% CI 2-sided [-2.09 to 1.07], Standard Error of Mean 0.80
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; Change in ADL UPDRS subscale of Isradipine CR 20mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.3674, ANCOVA; Mean Difference (Net) = -0.74, 95% CI 2-sided [-2.36 to 0.88], Standard Error of Mean 0.81

5. Secondary Outcome: Efficacy: Change in Motor Subscale of the Unified Parkinson's Disease Rating Scale
Description: The outcome is defined as change in Motor subscale of the Unified Parkinson's Disease Rating Scale(UPDRS Part III) between the baseline visit and month 12 or the time of sufficient disability to require dopaminergic therapy. UPDRS Part III: motor abilities at the time of the visit, consisting of 27 items (including 13 general questions and 14 sub-questions) each answered on a 0-4 point scale where 0 represents the absence of impairment and 4 represents the highest degree of impairment. Total Part III score represents the sum of these 27 items. A total of 108 points are possible. 108 represents the worst (total) disability), 0--no disability.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Population: All participants were included in primary and secondary outcome analyses
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
units on a scale | 4.32 (1.03) | 3.49 (1.09) | 3.91 (1.03) | 3.69 (1.07)
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; Change in Motor UPDRS subscale of Isradipine CR 5mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.579, ANCOVA; Mean Difference (Net) = -0.83, 95% CI 2-sided [-3.80 to 2.14], Standard Error of Mean 1.50
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; Change in Motor UPDRS subscale of Isradipine CR 10mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.7778, ANCOVA; Mean Difference (Net) = -0.41, 95% CI 2-sided [-3.30 to 2.48], Standard Error of Mean 1.46
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; Change in Motor UPDRS subscale of Isradipine CR 20mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.669, ANCOVA; Mean Difference (Net) = -0.64, 95% CI 2-sided [-3.58 to 2.31], Standard Error of Mean 1.48

6. Secondary Outcome: Efficacy: Change in Modified Hoehn & Yahr Scale
Description: The Modified Hoehn & Yahr Scale is an 8-level Parkinson's disease staging instrument. The outcome is defined as change in Modified Hoehn & Yahr Scale between the baseline visit and month 12 or the time of sufficient disability to require dopaminergic therapy. A greater increase in stage indicates a greater increase in disability. Stage ranges from 0-5 (also including 1.5 and 2.5) with 0 indicating no disability and 5 indicating maximum disability.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Population: All participants were included in primary and secondary outcome analyses
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
units on a scale | 0.27 (0.08) | 0.22 (0.08) | 0.12 (0.08) | 0.11 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; Change in Modified Hoehn & Yahr Scale of Isradipine CR 5mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.6677, ANCOVA; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.27 to 0.17], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; Change in Modified Hoehn & Yahr Scale of Isradipine CR 10mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.1755, ANCOVA; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.36 to 0.07], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; Change in Modified Hoehn & Yahr Scale of Isradipine CR 20mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.1463, ANCOVA; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.38 to 0.06], Standard Error of Mean 0.11

7. Secondary Outcome: Efficacy: Change in Modified Schwab & England Independence Scale
Description: The Schwab & England scale is an investigator and subject assessment of the subject's level of independence at all scheduled study visits. The subject will be scored on a percentage scale reflective of his/her ability to perform acts of daily living in relation to what he/she did before Parkinson's disease appeared. The outcome is defined as change in Schwab & England Independence Scale between the baseline visit and month 12 or the time of sufficient disability to require dopaminergic therapy. Higher decrease in score indicates higher disability. Score ranges from 100% (complete independence) to 0% (total disability).
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Population: All participants were included in primary and secondary outcome analyses
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
units on a scale | -5.04 (0.96) | -5.56 (1.02) | -3.69 (0.96) | -3.76 (1.01)
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; Change in Modified Schwab & England Independence Scale of Isradipine CR 5mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.7111, ANCOVA; Mean Difference (Net) = -0.52, 95% CI 2-sided [-3.30 to 2.26], Standard Error of Mean 1.40
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; Change in Modified Schwab & England Independence Scale of Isradipine CR 10mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.3237, ANCOVA; Mean Difference (Net) = 1.35, 95% CI 2-sided [-1.35 to 4.04], Standard Error of Mean 1.36
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; Change in Modified Schwab & England Independence Scale of Isradipine CR 20mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.3658, ANCOVA; Mean Difference (Net) = 1.27, 95% CI 2-sided [-1.51 to 4.05], Standard Error of Mean 1.40

8. Secondary Outcome: Efficacy: Change in Beck Depression Inventory II (BDI-II)
Description: The Beck Depression Inventory (BDI) is a validated self-reported 21-item depression scale that was tested and validated as a reliable instrument for screening for depression in PD. The outcome is defined as change in BDI-II between the baseline visit and month 12 or the time of sufficient disability to require dopaminergic therapy. Total BDI score represents the sum of these 21-items. A higher change in score indicates a greater increase in disability. Total score of 0-13 is considered minimal, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Population: All participants were included in primary and secondary outcome analyses
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
units on a scale | -0.52 (0.93) | 1.99 (0.93) | 0.11 (0.98) | 1.50 (0.95)
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; Change in BDI-II of Isradipine CR 5mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.0608, ANCOVA; Mean Difference (Net) = 2.50, 95% CI 2-sided [-0.12 to 5.13], Standard Error of Mean 1.32
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; Change in BDI-II of Isradipine CR 10mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.6445, ANCOVA; Mean Difference (Net) = 0.63, 95% CI 2-sided [-2.07 to 3.33], Standard Error of Mean 1.36
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; Change in BDI-II of Isradipine CR 20mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.1336, ANCOVA; Mean Difference (Net) = 2.02, 95% CI 2-sided [-0.63 to 4.67], Standard Error of Mean 1.52

9. Secondary Outcome: Efficacy: Change in Montreal Cognitive Assessment
Description: The Montreal Cognitive Assessment(MoCA) is a brief 30-point screening instrument that was developed and validated to identify subjects with mild cognitive impairment. The outcome is defined as change in MoCA between the baseline visit and month 12 or the time of sufficient disability to require dopaminergic therapy. Total MoCA score represents the sum of these 30-points, with a lower score indicating greater cognitive impairment. 30 is the maximum score, with a score of 26 or higher considered normal and below 26 indicative of Mild Cognitive Impairment.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Population: All participants were included in primary and secondary outcome analyses
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
units on a scale | 0.58 (0.40) | 0.06 (0.38) | 0.11 (0.41) | 0.36 (0.40)
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; Change in Montreal Cognitive Assessment of Isradipine CR 5mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.3533, ANCOVA; Mean Difference (Net) = -0.52, 95% CI 2-sided [-1.64 to 0.59], Standard Error of Mean 0.56
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; Change in Montreal Cognitive Assessment of Isradipine CR 10mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.4045, ANCOVA; Mean Difference (Net) = -0.47, 95% CI 2-sided [-1.59 to 0.65], Standard Error of Mean 0.56
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; Change in Montreal Cognitive Assessment of Isradipine CR 20mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.7049, ANCOVA; Mean Difference (Net) = -0.22, 95% CI 2-sided [-1.36 to 0.92], Standard Error of Mean 0.57

10. Secondary Outcome: Efficacy: Change in Parkinson Disease Quality of Life Questionnaire-39(PDQ-39)
Description: The PD Quality of Life Scale(PDQ-39) asks the subject to evaluate how Parkinson disease has affected their health and overall quality of life at that point in time. The total quality of life scale includes subscales relating to social role, self-image/sexuality, sleep, outlook, physical function and urinary function. The outcome is defined as change in PDQ-39 between the baseline visit and month 12 or the time of sufficient disability to require dopaminergic therapy. It is scored on a scale of zero to 100, with lower scores indicating better health and higher scores more severe disability.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Population: All participants were included in primary and secondary outcome analyses
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
units on a scale | 1.28 (1.28) | 3.47 (1.27) | 3.00 (1.35) | 3.35 (1.31)
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; Change in PDQ-39 of Isradipine CR 5mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.2278, ANCOVA; Mean Difference (Net) = 2.19, 95% CI 2-sided [-1.40 to 5.79], Standard Error of Mean 1.80
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; Change in PDQ-39 of Isradipine CR 5mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.356, ANCOVA; Mean Difference (Net) = 1.72, 95% CI 2-sided [-1.97 to 5.42], Standard Error of Mean 1.86
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; Change in PDQ-39 of Isradipine CR 20mg/day arm is compared to placebo group; Test type: Superiority or Other; p = 0.2600, ANCOVA; Mean Difference (Net) = 2.07, 95% CI 2-sided [-1.56 to 5.71], Standard Error of Mean 1.83

11. Secondary Outcome: Vital Signs: Change in Systolic Standing
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
mm Hg | -4.77 (2.49) | -9.85 (2.71) | -7.75 (2.60) | -6.30 (2.94)

12. Secondary Outcome: Vital Signs: Change in Systolic Supine
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
mm Hg | -2.45 (2.25) | -8.59 (2.45) | -6.45 (2.34) | -7.01 (2.65)

13. Secondary Outcome: Vital Signs: Change in Diastolic Standing
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
mm Hg | -0.38 (1.44) | -4.20 (1.57) | -5.14 (1.50) | -4.34 (1.69)

14. Secondary Outcome: Vital Signs: Change in Diastolic Supine
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
mm Hg | 0.09 (1.27) | -2.79 (1.38) | -4.54 (1.32) | -3.63 (1.49)

15. Secondary Outcome: Vital Signs: Change in Pulse Standing
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
beats per minute | -0.08 (1.89) | -2.98 (2.07) | -2.29 (1.97) | -1.21 (2.23)

16. Secondary Outcome: Vital Signs: Change in Pulse Supine
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
beats per minute | -0.42 (1.55) | -0.71 (1.69) | -0.52 (1.62) | 0.18 (1.83)

17. Secondary Outcome: Common Adverse Events: Oedema Peripheral
Description: General disorders and administration site conditions. Common adverse experience/event is defined as AE occurs to 5(about 5%) or more subjects.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 1 | 4 | 10 | 16
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; The analyses is to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Oedema Peripheral; Test type: Superiority or Other; p = 0.1384, Fisher Exact — The analysis of common AE of each active dosage of isradipine CR will be compared with that of the placebo group using one-sided Fisher's exact tests. No adjustment will be made for multiple comparisons in these analyses; Odds Ratio (OR) = 5.2632, 95% CI 2-sided [0.5432 to 50.9977], Standard Error of Mean 1.159
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Oedema Peripheral; Test type: Superiority or Other; p = 0.0024, Fisher Exact — [p-value comment as in outcome 17, analysis 1]; Odds Ratio (OR) = 15.6250, 95% CI 2-sided [1.8214 to 134.0403], Standard Error of Mean 1.097
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; Fisher's exact test will be used to compare Isradipine CR 20mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Oedema Peripheral; Test type: Superiority or Other; p < .0001, Fisher Exact — [p-value comment as in outcome 17, analysis 1]; Odds Ratio (OR) = 50.0000, 95% CI 2-sided [5.7004 to 438.5694], Standard Error of Mean 1.108

18. Secondary Outcome: Common Adverse Events: Dizziness
Description: Nervous system disorders. Common adverse experience/event is defined as AE occurs to 5(about 5%) or more subjects. They will also be tabulated by treatment groups.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 7 | 5 | 6 | 6
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; one-sided Fisher's exact test will be used to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Dizziness; Test type: Superiority or Other; p = 0.7735, Fisher Exact; Odds Ratio (OR) = 0.7540, 95% CI 2-sided [0.2022 to 2.8120], Standard Error of Mean 0.6715
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; one-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Dizziness; Test type: Superiority or Other; p = 0.7385, Fisher Exact; Odds Ratio (OR) = 0.8143, 95% CI 2-sided [0.2314 to 2.8658], Standard Error of Mean 0.6419
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 20mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Dizziness; Test type: Superiority or Other; p = 0.6823, Fisher Exact; Odds Ratio (OR) = 0.9048, 95% CI 2-sided [0.2549 to 3.2112], Standard Error of Mean 0.6463

19. Secondary Outcome: Common Adverse Events: Nasopharyngitis
Description: Infections and infestations. Common adverse experience/event is defined as AE occurs to 5(about 5%) or more subjects. They will also be tabulated by treatment groups.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 2 | 4 | 7 | 4
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Nasopharyngitis; Test type: Superiority or Other; p = 0.2756, Fisher Exact; Odds Ratio (OR) = 2.5263, 95% CI 2-sided [0.4172 to 15.2975], Standard Error of Mean 0.9188
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Nasopharyngitis; Test type: Superiority or Other; p = 0.07, Fisher Exact; Odds Ratio (OR) = 4.4211, 95% CI 2-sided [0.8217 to 23.7875], Standard Error of Mean 0.8584
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 20mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Nasopharyngitis; Test type: Superiority or Other; p = 0.2953, Fisher Exact; Odds Ratio (OR) = 2.4000, 95% CI 2-sided [0.3975 to 14.4919], Standard Error of Mean 0.9174

20. Secondary Outcome: Common Adverse Events: Headache
Description: as for outcome 18
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 3 | 3 | 6 | 4
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Headache; Test type: Superiority or Other; p = 0.6049, Fisher Exact; Odds Ratio (OR) = 1.1500, 95% CI 2-sided [0.2082 to 6.3508], Standard Error of Mean 0.8719
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Headache; Test type: Superiority or Other; p = 0.2327, Fisher Exact; Odds Ratio (OR) = 2.3000, 95% CI 2-sided [0.5081 to 10.4105], Standard Error of Mean 0.7704
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 20mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Headache; Test type: Superiority or Other; p = 0.4534, Fisher Exact; Odds Ratio (OR) = 1.5333, 95% CI 2-sided [0.3057 to 7.6897], Standard Error of Mean 0.8227

21. Secondary Outcome: Common Adverse Events: Constipation
Description: Gastrointestinal Disorders. Common adverse experience/event is defined as AE occurs to 5(about 5%) or more subjects. They will also be tabulated by treatment groups.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 3 | 2 | 3 | 4
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Constipation; Test type: Superiority or Other; p = 0.7852, Fisher Exact; Odds Ratio (OR) = 0.7302, 95% CI 2-sided [0.1109 to 4.8065], Standard Error of Mean 0.9616
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Constipation; Test type: Superiority or Other; p = 0.666, Fisher Exact; Odds Ratio (OR) = 1.0000, 95% CI 2-sided [0.1824 to 5.4820], Standard Error of Mean 0.8681
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 20mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Constipation; Test type: Superiority or Other; p = 0.4534, Fisher Exact; Odds Ratio (OR) = 1.5333, 95% CI 2-sided [0.3057 to 7.6897], Standard Error of Mean 0.8227

22. Secondary Outcome: Common Adverse Events: Fatigue
Description: General Disorders and Administration Site Conditions. Common adverse experience/event is defined as AE occurs to 5(about 5%) or more subjects. They will also be tabulated by treatment groups.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 2 | 1 | 3 | 3
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Fatigue; Test type: Superiority or Other; p = 0.8589, Fisher Exact; Odds Ratio (OR) = 0.5455, 95% CI 2-sided [0.0462 to 6.4433], Standard Error of Mean 1.2596
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Fatigue; Test type: Superiority or Other; p = 0.5000, Fisher Exact; Odds Ratio (OR) = 1.5652, 95% CI 2-sided [0.2392 to 10.2410], Standard Error of Mean 0.9584
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 20mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Fatigue; Test type: Superiority or Other; p = 0.4609, Fisher Exact; Odds Ratio (OR) = 1.7143, 95% CI 2-sided [0.2609 to 11.2639], Standard Error of Mean 0.9605

23. Secondary Outcome: Common Adverse Events: Nausea
Description: as for outcome 21
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 3 | 2 | 1 | 2
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Nausea; Test type: Superiority or Other; p = 0.7852, Fisher Exact; Odds Ratio (OR) = 0.7302, 95% CI 2-sided [0.1109 to 4.8065], Standard Error of Mean 0.9616
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Nausea; Test type: Superiority or Other; p = 0.9448, Fisher Exact; Odds Ratio (OR) = 0.3067, 95% CI 2-sided [0.0297 to 3.1612], Standard Error of Mean 1.1912
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 20mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Nausea; Test type: Superiority or Other; p = 0.7996, Fisher Exact; Odds Ratio (OR) = 0.6970, 95% CI 2-sided [0.1061 to 4.5779], Standard Error of Mean 0.9604

24. Secondary Outcome: Common Adverse Events: Upper Respiratory Tract Infection
Description: as for outcome 19
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 1 | 2 | 5 | 0
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Tract Infection; Test type: Superiority or Other; p = 0.4532, Fisher Exact; Odds Ratio (OR) = 2.3810, 95% CI 2-sided [0.2015 to 28.1366], Standard Error of Mean 1.2599
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Tract Infection; Test type: Superiority or Other; p = 0.0953, Fisher Exact; Odds Ratio (OR) = 5.9524, 95% CI 2-sided [0.6439 to 55.0272], Standard Error of Mean 1.1347

25. Secondary Outcome: Common Adverse Events: Depression
Description: Psychiatric Disorders. Common adverse experience/event is defined as AE occurs to 5(about 5%) or more subjects. They will also be tabulated by treatment groups.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 2 | 3 | 1 | 1
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Depression; Test type: Superiority or Other; p = 0.4402, Fisher Exact; Odds Ratio (OR) = 1.8000, 95% CI [0.2733 to 11.8558], Standard Error of Mean 0.9617
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Depression; Test type: Superiority or Other; p = 0.8824, Fisher Exact; Odds Ratio (OR) = 0.4800, 95% CI 2-sided [0.0408 to 5.6461], Standard Error of Mean 1.2577
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 20mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Depression; Test type: Superiority or Other; p = 0.6641, Fisher Exact; Odds Ratio (OR) = 1.0909, 95% CI 2-sided [0.1413 to 8.4197], Standard Error of Mean 1.0428

26. Secondary Outcome: Common Adverse Events: Somnolence
Description: as for outcome 18
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 2 | 3 | 2 | 0
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Somnolence; Test type: Superiority or Other; p = 0.4402, Fisher Exact; Odds Ratio (OR) = 1.8000, 95% CI 2-sided [0.2733 to 11.8558], Standard Error of Mean 0.9617
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Somnolence; Test type: Superiority or Other; p = 0.6951, Fisher Exact; Odds Ratio (OR) = 1.0000, 95% CI 2-sided [0.1300 to 7.6906], Standard Error of Mean 1.0409

27. Secondary Outcome: Common Adverse Events: Insomnia
Description: as for outcome 25
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 2 | 3 | 1 | 1
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Insomnia; Test type: Superiority or Other; p = 0.4402, Fisher Exact; Odds Ratio (OR) = 1.8000, 95% CI 2-sided [0.2733 to 11.8558], Standard Error of Mean 0.9617
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Insomnia; Test type: Superiority or Other; p = 0.8824, Fisher Exact; Odds Ratio (OR) = 0.4800, 95% CI 2-sided [0.0408 to 5.6461], Standard Error of Mean 1.2577
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 20mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Insomnia; Test type: Superiority or Other; p = 0.8673, Fisher Exact; Odds Ratio (OR) = 0.5217, 95% CI 2-sided [0.0442 to 6.1537], Standard Error of Mean 1.2594

28. Secondary Outcome: Common Adverse Events: Dyspepsia
Description: as for outcome 21
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 3 | 1 | 1 | 1
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Dyspepsia; Test type: Superiority or Other; p = 0.9294, Fisher Exact; Odds Ratio (OR) = 0.3485, 95% CI 2-sided [0.0337 to 3.6084], Standard Error of Mean 1.1919
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Dyspepsia; Test type: Superiority or Other; p = 0.9448, Fisher Exact; Odds Ratio (OR) = 0.3067, 95% CI 2-sided [0.0297 to 3.1612], Standard Error of Mean 1.1912
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 20mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Dyspepsia; Test type: Superiority or Other; p = 0.9351, Fisher Exact; Odds Ratio (OR) = 0.3333, 95% CI 2-sided [0.0322 to 3.4459], Standard Error of Mean 1.1924

29. Secondary Outcome: Common Adverse Events: Diarrhoea
Description: as for outcome 21
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 2 | 1 | 2 | 1
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Diarrhoea; Test type: Superiority or Other; p = 0.8589, Fisher Exact; Odds Ratio (OR) = 0.5455, 95% CI 2-sided [0.0462 to 6.4433], Standard Error of Mean 1.2596
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Diarrhoea; Test type: Superiority or Other; p = 0.6951, Fisher Exact; Odds Ratio (OR) = 1.0000, 95% CI 2-sided [0.1300 to 7.6906], Standard Error of Mean 1.0409
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 20mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Diarrhoea; Test type: Superiority or Other; p = 0.8673, Fisher Exact; Odds Ratio (OR) = 0.5217, 95% CI 2-sided [0.0442 to 6.1537], Standard Error of Mean 1.2594

30. Secondary Outcome: Common Adverse Events: Sinusitis
Description: as for outcome 19
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 3 | 2 | 1 | 0
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Sinusitis; Test type: Superiority or Other; p = 0.7852, Fisher Exact; Odds Ratio (OR) = 0.7302, 95% CI 2-sided [0.1109 to 4.8065], Standard Error of Mean 0.9616
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Sinusitis; Test type: Superiority or Other; p = 0.9448, Fisher Exact; Odds Ratio (OR) = 0.3067, 95% CI 2-sided [0.0297 to 3.1612], Standard Error of Mean 1.1912

31. Secondary Outcome: Common Adverse Events: Back Pain
Description: Musculoskeletal and Connective Tissue Disorders. Common adverse experience/event is defined as AE occurs to 5(about 5%) or more subjects. They will also be tabulated by treatment groups.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 1 | 0 | 2 | 3
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 10mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Back Pain; Test type: Superiority or Other; p = 0.5000, Fisher Exact; Odds Ratio (OR) = 2.0833, 95% CI 2-sided [0.1771 to 24.5057], Standard Error of Mean 1.2576
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 20mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 20mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Back Pain; Test type: Superiority or Other; p = 0.2746, Fisher Exact; Odds Ratio (OR) = 3.5714, 95% CI 2-sided [0.3453 to 36.9408], Standard Error of Mean 1.192

32. Secondary Outcome: Common Adverse Events: Hypotension
Description: Vascular Disorders. Common adverse experience/event is defined as AE occurs to 5(about 5%) or more subjects. They will also be tabulated by treatment groups.
Time Frame: Baseline to 12 months or the time to require dopaminergic therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Number analyzed (Participants) | 26 | 23 | 26 | 24
participants | 1 | 1 | 2 | 2
Statistical Analysis 1: Comparison: Placebo vs Isradipine CR 5mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 5mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Hypotension; Test type: Superiority or Other; p = 0.7236, Fisher Exact; Odds Ratio (OR) = 1.1364, 95% CI 2-sided [0.0670 to 19.2640], Standard Error of Mean 1.4444
Statistical Analysis 2: Comparison: Placebo vs Isradipine CR 10mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 10mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Hypotension; Test type: Superiority or Other; p = 0.5000, Fisher Exact; Odds Ratio (OR) = 2.0833, 95% CI 2-sided [0.1771 to 24.5057], Standard Error of Mean 1.2576
Statistical Analysis 3: Comparison: Placebo vs Isradipine CR 20mg/Day; One-sided Fisher's exact test will be used to compare Isradipine CR 20mg group to the placebo group with regard to the proportion of subjects experiencing the adverse event of Hypotension; Test type: Superiority or Other; p = 0.4694, Fisher Exact; Odds Ratio (OR) = 2.2727, 95% CI 2-sided [0.1926 to 26.8124], Standard Error of Mean 1.2592

ADVERSE EVENTS:
Time Frame: 12 months or the time to require dopaminergic therapy
Description: All serious and most common adverse experiences/events will be listed by treatment. Most common adverse experiences/events were defined as AEs occurring more than 5 times(5%).
Arm/Group | Placebo | Isradipine CR 5mg/Day | Isradipine CR 10mg/Day | Isradipine CR 20mg/Day
Serious Adverse Events (participants affected / at risk) | 2/26 | 2/23 | 1/26 | 2/24
Other Adverse Events (participants affected / at risk) | 23/26 | 21/23 | 23/26 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | Isradipine CR 5mg/Day (N=23) | Isradipine CR 10mg/Day (N=26) | Isradipine CR 20mg/Day (N=24)
PYREXIA (General disorders) | 0 | 1 | 0 | 0
VITRECTOMY (Surgical and medical procedures) | 1 | 0 | 0 | 0
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 1 | 0 | 0 — Subject #5222
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 0 | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | Isradipine CR 5mg/Day (N=23) | Isradipine CR 10mg/Day (N=26) | Isradipine CR 20mg/Day (N=24)
Oedema Peripheral (General disorders) | 1 | 4 | 10 | 16
Dizziness (Nervous system disorders) | 7 | 5 | 6 | 6
Nasopharyngitis (Infections and infestations) | 2 | 4 | 7 | 4
Headache (Nervous system disorders) | 3 | 3 | 6 | 4
Constipation (Gastrointestinal disorders) | 3 | 2 | 3 | 4
Fatigue (General disorders) | 2 | 1 | 3 | 3
Nausea (Gastrointestinal disorders) | 3 | 2 | 1 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 5 | 0
Depression (Psychiatric disorders) | 2 | 3 | 1 | 1
Somnolence (Nervous system disorders) | 2 | 3 | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 3 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2 | 1
Sinusitis (Infections and infestations) | 3 | 2 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3
Hypotension (Vascular disorders) | 1 | 1 | 2 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No